CLINICAL TRIAL: NCT04635358
Title: Feasibility Study of Smoking Cessation for the Staff of a Hospital Center Through a Treatment Proposal Combining Nicotine Substitutes, Psychological Support, Nutritional Assistance and Hypnosis.
Brief Title: Feasibility Study of Smoking Cessation for the Staff of a Hospital Center
Acronym: Je_Respire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-PP-16
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Smoking Cessation
Keywords: Smoking, hypnosis, nutrition support, psychological support
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Setting up hypnosis sessions, psychological and nutritional assistance.
  Interventions: Behavioral: Hypnosis; Behavioral: Psychological support; Behavioral: Nutrional support

INTERVENTIONS:
Behavioral: Hypnosis — Setting up hypnosis sessions
Behavioral: Psychological support — Setting up psychological support
Behavioral: Nutrional support — Setting up nutritional support

SUMMARY:
The recorded prevalence of daily smoking among health professionals (doctors, nurses, midwives, etc.), regardless of their mode of practice (salaried or self-employed, etc.) varies between 14 and 23%. In health care institutions, according to the studies, the prevalence of daily smoking among staff, caregivers and non-caregivers ranges from 17% to 27%. These professionals who continue to smoke, although they are particularly well informed about the risks they run, probably constitute a group with specific withdrawal difficulties. Beyond the impact on their own health, the smoking status of caregivers could also have an impact on the management of tobacco patients. There are very few studies of the impact of interventions on the smoking status of caregivers in health care facilities. The combination of several intervention modalities can facilitate the participation of target professionals and generate efficiency synergies.

ELIGIBILITY:
Inclusion Criteria:

Professionals employed at the Nice hospital who are volunteers and have :

* an initial Fagerstrom test > 3
* associated with expired carbone monoxide > 10 ppm at least 60' after the last cigarette.

Exclusion Criteria:

* Reported associated addiction (cannabis, alcohol or any other psychoactive product)
* Professionals likely to no longer work at the Nice Hospital in the year following the start of the study
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects enrolled in the program who participated in the full range of care offered | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard PROUVOST-KELLER, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No